CLINICAL TRIAL: NCT03037658
Title: Physical Activity Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Laura L Carstensen, Professor of Psychology and the Fairleigh S. Dickinson Jr. Professor in Public Policy, Director of the Stanford Center on Longevity, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-28280
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Physical Activity
Keywords: physical activity; walking; incentive; step count
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Personal - self (Experimental): Participants had the opportunity to earn money for themselves by increasing their average steps per day.
  Interventions: Other: Offering a financial incentive to increase walking
- Prosocial - loved one (Experimental): Participants had the opportunity to earn money for a loved one of their choice by increasing their average steps per day.
  Interventions: Other: Offering a financial incentive to increase walking
- Prosocial - charity (Experimental): Participants had the opportunity to earn money for a charity of their choice by increasing their average steps per day.
  Interventions: Other: Offering a financial incentive to increase walking
- Choice (Experimental): Participants were given the choice to earn money either for themselves, a loved one, or a charity by increasing their average steps per day.
  Interventions: Other: Offering a financial incentive to increase walking
- Control (No Intervention): Participants were not offered a financial incentive to increase their average steps per day. They simply wore the pedometer for three weeks.

INTERVENTIONS:
Other: Offering a financial incentive to increase walking — After a baseline week of walking while wearing a pedometer, participants will be randomly assigned to one of the five conditions. In each of these conditions, participants will have the chance to earn .02/step for each additional step per day (on average across the week, above baseline levels). After a week of incentivized walking, participants will again be asked to wear the pedometer for one final week (with no incentive).
  Because the investigators need a week of walking before the incentive week, it is important that participants do not know the specific incentive aspect at the beginning of the study. Therefore, the investigators will not disclose the incentive structure at the beginning of the study. The investigators will debrief participants at the end of the study, and they will be fully informed of the purposes of the study at that time.
  Arms: Choice; Personal - self; Prosocial - charity; Prosocial - loved one

SUMMARY:
In this study, the investigators will test responsiveness of young, middle-aged, and older adults to a range of incentives, some of which provide rewards for the individual participants and others that offer rewards to other people or groups. The investigators hypothesize that incentives are differentially effective for different age groups.

DETAILED DESCRIPTION:
This study grounds a financial incentives intervention in well-documented age-related changes in motivation. The investigators consider these motivational shifts through the lens of socioemotional selectivity theory (SST, Carstensen, 2006). According to SST, perceived time horizons influence motivation across the life span. When time is perceived as expansive (typical of younger adults), exploration and achievement are prioritized, but when time horizons narrow (typical of older adults), emotional meaning and satisfaction are prioritized. Previous research has shown that socioemotional goals may influence decisions about healthcare plans and the effectiveness of motivational messages to increase physical activity (Löckenhoff & Carstensen, 2007; Mikels et al., 2010; Notthoff & Carstensen, 2013). Drawing on the tenets of SST, individuals may be more motivated to engage in physical activity when doing so aligns with socioemotional goals. For example, older adults may find physical activity most appealing when it promotes emotional meaning and satisfaction; in contrast, younger adults may find physical activity most appealing when it promotes exploration and achievement.

Recent work has shown that spending on others (termed "prosocial spending") can have greater emotional benefits than spending on oneself (Anik, Aknin, Norton, Dunn, & Quoidbach, 2013; Dunn, Aknin, & Norton, 2008). Extending this concept, the researchers posit that, in the context of financial incentives, earning for others may offer older adults a more emotionally meaningful alternative to individual financial incentives, which may, in turn, better support health behavior change for older adults. Because of the profound link between physical activity and risk for cardiovascular disease and stroke, and because previous research suggests that financial incentives are most effective for simple, well-defined, objectively measurable activities, the behavioral outcome of interest in this study focuses on walking measured by pedometer step counts (Scott & Schurer, 2008). In addition, because SST postulates specifically about motivational priorities in younger relative to older adults, the investigators recruited adult participants of all ages. The researchers designed this study to test the effectiveness of prosocial relative to individual financial incentives for increasing walking in older and younger adults. Reasoning from SST, the investigators hypothesize that younger adults will be relatively more motivated by incentives that produce personal benefits (i.e. individual financial incentives), but older adults will be relatively more affected when incentives were more emotionally meaningful (i.e. benefit another person or social cause). The investigators also predict that, when given the choice of incentive, older adults will be more likely to choose to earn for others rather than to earn for themselves, relative to younger adults. In addition, the investigators will also test the effects of prosocial relative to individual financial incentives on intrinsic motivation for physical activity and behavioral maintenance (maintaining increased steps) once incentives are removed.

Community-residing adults aged 18 and older are recruited via advertisements on Internet bulletin boards and local newspapers to participate in a study that requires four visits to our laboratory and three weeks of pedometer wear in exchange for $50. Importantly, participants are unaware of the incentive component of this study. Once participants contact research staff to indicate their interest, they are phone screened for eligibility (see the eligibility criteria section of this entry).

During the first in-lab session, after providing informed consent, participants respond to a series of questionnaires using Qualtrics survey software. Participants are provided with a pedometer, instructed on its use, and asked to wear it each day. One week later, participants return to complete the second study session. Participants complete questionnaires while pedometer steps are downloaded. Participants are randomly assigned within age group and gender to one of five possible incentive conditions (which can be found in the arms and interventions section of this entry). One week later, participants return to the lab for the third study session where they complete questionnaires while pedometer steps are downloaded. All participants are told their average daily steps from the previous week and how this average relates to the first week's average. Participants in incentivized conditions who increase steps are told how much they earned. Participants in the personal condition and choice participants who elect to keep the earnings receive a check for the amount of their earnings. Participants in the loved one and charity conditions and choice participants who elect to give their earnings to a loved one or charity witness the research staff write a check for the amount of their earnings to their selected loved one or charity and enclose the check along with a cover letter into an envelope to be mailed. Participants in the incentivized conditions who do not increase steps were told that they did not earn any money. All participants in incentivized conditions are reminded that the incentive portion of the study is complete and that they will not earn money by changing steps the final week of the study. One week later, participants complete the final study session. Participants complete questionnaires while pedometer steps are downloaded. All participants are told their average daily steps from the previous week and how this average relates to the second week's average. At the end of the session, participants are debriefed, paid, and thanked for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older are being targeted. We aim to recruit equal numbers of men and women, but this is not a specific target. There are no racial or ethnic targets.
* Individuals who pass a phone screening that includes physical (PAR-Q) and cognitive (MMSE) measures are eligible for this study. These individuals must either answer "no" to all the questions on the Physical Activity Readiness Questionnaire (PAR-Q) or receive verbal permission from their doctor. Additionally, they must also show no signs of cognitive impairment as indicated by scores greater than or equal to 23 points on the 26-point Mini-Mental State Examination (MMSE).

Exclusion Criteria:

* We will not recruit minors (17 or younger) because this is a study of adult development.
* Individuals who answered "yes" on any questions of the PAR-Q and/or received a score less than or equal to 22 on the MMSE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in average steps per day | Step count is measured via pedometer every day for three weeks
  Difference in average steps per day (from baseline week to incentive week)

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Carstensen, PhD, Principal Investigator — Stanford University
Locations (1):
- Life-span Development Lab, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers will share de-identified participant data with other researchers.

REFERENCES:
- [Background] Carstensen LL. The influence of a sense of time on human development. Science. 2006 Jun 30;312(5782):1913-5. doi: 10.1126/science.1127488. PMID 16809530
- [Background] Lockenhoff CE, Carstensen LL. Aging, emotion, and health-related decision strategies: motivational manipulations can reduce age differences. Psychol Aging. 2007 Mar;22(1):134-146. doi: 10.1037/0882-7974.22.1.134. PMID 17385990
- [Background] Mikels JA, Lockenhoff CE, Maglio SJ, Goldstein MK, Garber A, Carstensen LL. Following your heart or your head: focusing on emotions versus information differentially influences the decisions of younger and older adults. J Exp Psychol Appl. 2010 Mar;16(1):87-95. doi: 10.1037/a0018500. PMID 20350046
- [Background] Notthoff N, Carstensen LL. Positive messaging promotes walking in older adults. Psychol Aging. 2014 Jun;29(2):329-341. doi: 10.1037/a0036748. PMID 24956001
- [Background] Anik L, Aknin LB, Norton MI, Dunn EW, Quoidbach J. Prosocial bonuses increase employee satisfaction and team performance. PLoS One. 2013 Sep 18;8(9):e75509. doi: 10.1371/journal.pone.0075509. eCollection 2013. PMID 24058691
- [Background] Dunn EW, Aknin LB, Norton MI. Spending money on others promotes happiness. Science. 2008 Mar 21;319(5870):1687-8. doi: 10.1126/science.1150952. PMID 18356530
- [Background] Scott A, Schurer S. Financial incentives, personal responsibility and prevention. Discussion paper comissioned by the National Health and Hospitals Reform Commission. 2008. Retrieved from: http://www.health.gov.au/internet/nhhrc/publishing.nsf/Content/discussion-papers
- [Derived] Raposo S, Hogan CL, Barnes JT, Chemudupati T, Carstensen LL. Leveraging goals to incentivize healthful behaviors across adulthood. Psychol Aging. 2021 Feb;36(1):57-68. doi: 10.1037/pag0000428. Epub 2020 Jul 6. PMID 32628030